CLINICAL TRIAL: NCT07245108
Title: The ProChol Study - Prospective Assessment of Symptoms Following Cholecystectomy in Patients With Symptomatic Uncomplicated Gallstones
Brief Title: The Pro-Chol Study
Acronym: ProChol
Status: Recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Hvidovre University Hospital (Other); Copenhagen University Hospital at Herlev (Other); Aalborg University Hospital (Other); Viborg Regional Hospital (Other); Zealand University Hospital (Other); University Hospital Bispebjerg and Frederiksberg (Other); Regionshospital Nordjylland (Other Government); Copenhagen University Hospital Nordsjælland (Unknown); Regionshospitalet Viborg, Skive (Other)
Responsible Party: Sponsor
Other Study IDs: P-2023-188
Record Dates: First submitted 2025-11-15; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Gallstones; Gallstone Attack; Uncomplicated Cholelithiasis; Cholecystolithiasis
Keywords: Cohort study; Prospective clinical study; Cholecystectomy; Laparoscopic cholecystectomy; Pain relief
MeSH Terms: conditions — Gallstones; Cholecystolithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with gallbladder stones and biliary pain that undergo laparoscopic cholecystectomy: Patients are included if they have gallbladder stones on abdominal ultrasound examination, abdominal pain expected to be due to gallstones by the clinician and scheduled for elective laparoscopic cholecystectomy. Patients with either a history including biliary interventions or complicated gallstone disease such as pancreatitis, cholecystitis or bile duct stones will be excluded.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — A surgical removal of the gallbladder through laparoscopy
Procedure: Laparoscopic cholecystectomy — The intervention is intended laparoscopic cholecystectomy. Patients that undergo conversion to open (traditional) cholecystectomy will still be included. Patients scheduled for open cholecystectomy will not be included.

SUMMARY:
This prospective clinical cohort study will include patients with gallstones and abdominal pain scheduled for surgery (laparoscopic cholecystectomy). Data on quality of life, abdominal pain, gallstone disease, and patient characteristics will be collected before surgery. The outcomes will be assessed three months following surgery and will primarily be determinants for resolution of pain. The aim is to make a prediction score that may aid clinicians and patients in decision making about surgery.

DETAILED DESCRIPTION:
Cholecystectomy is the surgical removal of the gallbladder and the only definitive treatment for both symptomatic complicated and uncomplicated gallstones. Surgery rates for laparoscopic cholecystectomy have been rapidly rising in European countries the past decades. Over 9000 cholecystectomies were performed in Denmark in 2016. Symptomatic outcomes following surgery have not been with the intended resolution of symptoms and remaining symptoms are reported in about 35% of patients. This indicates clinical challenges in selecting the patients that will benefit the most from surgery.

The quality of symptomatic outcomes following laparoscopic cholecystectomy should be assessed in a Danish population reflecting current clinical practice for selection of patients with symptomatic uncomplicated gallstones for surgery. Development of a clinical prediction tool for pain relief including both patient-reported and readily available objective variables could aid future patient selection and minimize overall health-care costs and unnecessary surgery risk in patients with symptomatic uncomplicated gallstones.

The aim is to perform a prospective assessment of the symptomatic outcomes of elective laparoscopic intended cholecystectomy in patients with symptomatic uncomplicated gallstones and to develop a prediction model for a pain-free state.

This is a prospective observational study that will be performed across the general surgical hospitals in healthcare regions of Denmark. Consecutive consenting patients will be included from each site until required sample size has reached.

Eligible patients will be identified through screening lists of outpatient clinics and of operating theaters. Patients will be approached for consent and data collection at either the outpatient clinical visit where cholecystectomy is scheduled or at a later timepoint before surgery. Follow-up for symptomatic outcome will be performed three months after surgery. Data collection at both study entry and follow-up will include access to the electronic patient record and answering an online patient questionnaire. If patient questionnaires remain unanswered after one week, the patient will be reminded through an online re-invitation. Data collection at entry will also include the patients' medical history and clinicopathological variables. Data will be stored in a purpose-build database in the clinical research platform REDCap.

The study will be run by a steering committee including senior surgeons acting as local investigators from each of the participating centers. The local investigator will ensure completion of data forms and follow-up procedures. An additional collaborator from each center may further be appointed responsible for patient identification and data collection.

This study is purely observational and no alterations to standard patient treatment will be performed.

A prediction model with high internal and external validity requires model development and validation to be performed in two independent sets of data. To ensure this, half of patients will be included for model development and the other half for model validation.

Based on a previous report, 60% (57%) will become pain-free following cholecystectomy. With a prediction model containing up to 12 exposure variables and a parameter to outcome event ratio of 1:20, the required sample size is 400 patients for model development. The total sample size will be 800 patients for both development and validation of the model. It is estimated that each center will identify about 20 eligible patients each month and the required inclusion period is therefore about two to three years. Sample size may be reduced if prediction model includes fewer variables.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound examination with presence of gallstones and description of size, number and presence of stones in infundibulum or cystic duct
* Abdominal symptoms believed to be caused by symptomatic uncomplicated gallstones
* Indication and candidate for elective laparoscopic cholecystectomy
* Above 18 years of age
* Ability to give oral and written consent
* Ability to understand, speak and read Danish
* Ability to receive digital post

Exclusion Criteria:

* History of complicated gallstone disease including acute cholecystitis, pancreatitis, common bile duct stones, or cholangitis
* Previous sphincterotomy
* Abnormal liver function test (ALAT/ASAT, alkaline phosphatase, bilirubin) without magnetic resonance cholangio-pancreatography or endoscopic ultrasound to rule out common bile duct pathology
* Indication for urgent cholecystectomy
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will include patients referred to outpatient clinics either from primary care general practitioners or from a hospital department. Currently six hospitals are included from four out of five Danish health care regions.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Prediction model for resolution of pain | From baseline before surgery to follow-up at three months after surgery
  To build and validate a prediction model for resolution of pain (VAS≤4) following laparoscopic cholecystectomy

SECONDARY OUTCOMES:
Changes in symptoms following surgery | From baseline before surgery to follow-up at three months after surgery
  To explore the changes in symptoms following cholecystectomy as defined through 1. core symptoms of the GIQLI questionnaire (such as dyspeptic symptoms, diarrhea, and constipation); 2. GIQLI quality of life total scores.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mønsted Shabanzadeh, DMSc, PhD, MD, Principal Investigator — Dansk: Offentligt hospital (inkl. universitetshospital)
Locations (7):
- Denmark (7):
  - Bispebjerg Hospital, Copenhagen, Bispebjerg
  - Aalborg Universitetshospital, Aalborg
  - Herlev Hospital, Herlev
  - Nordsjællands Hospital Hillerød, Hillerød
  - Regionshospital Nordjylland Hjørring, Hjørring
  - Hvidovre Hospital, Hvidovre
  - Regionshospital Viborg, Viborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Latenstein CSS, Hannink G, van der Bilt JDW, Donkervoort SC, Eijsbouts QAJ, Heisterkamp J, Nieuwenhuijs VB, Schreinemakers JMJ, Wiering B, Boermeester MA, Drenth JPH, van Laarhoven CJHM, Dijkgraaf MGW, de Reuver PR; SECURE trial collaborators. A Clinical Decision Tool for Selection of Patients With Symptomatic Cholelithiasis for Cholecystectomy Based on Reduction of Pain and a Pain-Free State Following Surgery. JAMA Surg. 2021 Oct 1;156(10):e213706. doi: 10.1001/jamasurg.2021.3706. Epub 2021 Oct 13. PMID 34379080
- [Background] Lamberts MP, Lugtenberg M, Rovers MM, Roukema AJ, Drenth JP, Westert GP, van Laarhoven CJ. Persistent and de novo symptoms after cholecystectomy: a systematic review of cholecystectomy effectiveness. Surg Endosc. 2013 Mar;27(3):709-18. doi: 10.1007/s00464-012-2516-9. Epub 2012 Oct 6. PMID 23052498
- [Background] Bray F, Balcaen T, Baro E, Gandon A, Ficheur G, Chazard E. Increased incidence of cholecystectomy related to gallbladder disease in France: Analysis of 807,307 cholecystectomy procedures over a period of seven years. J Visc Surg. 2019 Jun;156(3):209-215. doi: 10.1016/j.jviscsurg.2018.12.003. Epub 2018 Dec 18. PMID 30573436
- [Background] Lunevicius R, Nzenwa IC, Mesri M. A nationwide analysis of gallbladder surgery in England between 2000 and 2019. Surgery. 2022 Feb;171(2):276-284. doi: 10.1016/j.surg.2021.10.025. Epub 2021 Nov 12. PMID 34782153